CLINICAL TRIAL: NCT05230173
Title: Treat-to-Target of Endoscopic Remission in Patients With IBD in Symptomatic Remission
Acronym: QUOTIENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Baylor College of Medicine (Other); Crohn's and Colitis Foundation (Other); Western University (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Siddharth Singh, Associate Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RCT01519
Record Dates: First submitted 2022-01-27; First posted 2022-02-08 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Ulcerative Colitis; Crohn Disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease | interventions — Pragmatic Clinical Trials as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Switching Targeted Immunomodulators Treatment (Other): Participants randomized to a strategy of switching TIM will be switched to one of the preferred agents recommended by clinical guidelines and covered by the participants' insurance formulary as part of routine care, and at the discretion of the site investigator and treating provider. No study-related medications will be provided.
  For participants randomized to switch to an alternative TIM, selection of alternative agent will be determined at the discretion of the local site physician in accordance with clinical guidelines on the management of moderate to severe ulcerative colitis, and management of moderate to severe CD from the AGA and ACG.9, 34, 35 These guidelines include recommendations on positioning of TIMs for first line use (TIM-naïve patients) and second-line use (in patients with prior exposure to TIMs).
  Interventions: Other: Pragmatic
- Continuing Index Targeted Immunomodulators Treatment (Other): Participants randomized to a strategy of continuing TIM will continue on their concomitant therapy.
  Interventions: Other: Pragmatic

INTERVENTIONS:
Other: Pragmatic — Patients randomized to a strategy of switching TIM will be switched to one of the preferred agents recommended by clinical guidelines and covered by the patients' insurance formulary as part of routine care, and at the discretion of the site investigator and treating provider. No study-related medications will be provided.
  Patients (and their providers) in either treatment arm will be allowed to stop or start new TIMs and other IBD-directed therapies in case of symptomatic relapse or intolerance to therapies, at the discretion of the treating provider-patient team.

SUMMARY:
The purpose of this study is to compare the effectiveness and safety of a strategy of switching to an alternative targeted immunomodulator (TIM) therapy to treat to a target of endoscopic remission, versus continuing index TIM in patients with inflammatory bowel disease (IBD) (Crohn's disease or ulcerative colitis [UC]) in symptomatic remission with moderate to severe endoscopic inflammation despite optimization of index TIM in a real-world setting.

DETAILED DESCRIPTION:
This is a pragmatic, open-label, multicenter randomized control trial (RCT) conducted in asymptomatic patients with IBD who have persistent moderate to severe endoscopic inflammation despite optimization of index TIM. This study plans to recruit approximately 250 participants in the United States, who will either switching to treatment with alternative TIM to treat to a target of endoscopic remission or continue index optimized TIM. After randomization, patients will be followed prospectively within routine clinical practice over 2 years (104 weeks). This trial will be conducted within select active sites in the United States and Canada

The primary outcome will be time from randomization to treatment failure, as a composite of:

1. Moderate severe symptomatic relapse based on PRO2 (2-item patient reported outcome), with objective confirmation of inflammation within 2 months of event (fecal calprotectin [FC] >150 mcg/g, or C reactive protein [CRP] >5mg/L, or endoscopy showing moderate-severe inflammation, or magnetic resonance enterography (MRE)/computed tomography enterography (CTE)/intestinal ultrasound (IUS) showing active inflammation) with need for escalation of therapy;
2. Need for rescue therapy with corticosteroids for a documented symptomatic IBD flare;
3. IBD related hospitalization;
4. IBD-related surgery;
5. IBD-related structural complications (CD: symptomatic stricture, fistula or abscess; UC: symptomatic stricture);
6. Treatment-emergent adverse event requiring drug discontinuation.

Secondary outcomes will include time from randomization to each of the components in the primary outcome, quality of life (overall quality of life, fatigue, IBD-related disability), burden of treatment (financial burden, burden of monitoring, treatment side effects), treatment satisfaction, and safety.

In compliance with the pragmatic methodology of this study embedded in routine clinical care, there is no study visit mandated per study protocol. Participant visit schedules will follow local SOC with any additional visits at the treating physician's discretion. Data on all effectiveness, treatment burden and safety outcomes will be captured using a REDCap (Research Electronic Data Capture) database hosted at CCF. Data for the study will be extracted from medical record information and entered into the EDC system at baseline and then approximately every 6 months (at a minimum) thereafter, up to a 2-year follow-up period. Patient-reported outcome (PRO) measures (self-assessment questionnaires) will be utilized in this study to determine primary (efficacy) and secondary (quality of life and treatment burden and satisfaction) outcomes. Participants will complete the PRO2 at baseline and approximately every 12 weeks during a 2-year follow-up period; additional questionnaires (IBD-Control, PROMIS-7, Short Inflammatory Bowel Disease Questionnaire [SIBDQ], IBD Disability Index [IBD-DI], Treatment Burden Questionnaire, and Treatment Satisfaction Questionnaire for Medication) will be completed at baseline (following randomization) and up to 3 more additional times during a 2-year follow-up period.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Male or nonpregnant, nonlactating females, ≥ 18 years of age.
2. An established diagnosis of CD or UC for at least 6 months based on standard clinical criteria, confirmed by the treating provider.
3. Current treatment with an approved TIM for treatment of IBD, including biologic agents (e.g., TNFα antagonists, ustekinumab, vedolizumab) and small molecule inhibitors (e.g., Janus kinase inhibitors, ozanimod), including future TIMs that become commercially available during the conduct of the trial.
4. Dose of TIM should be stable for 3 or more months prior to qualifying endoscopy/radiology. No treatment escalation of TIM or addition of IMM, corticosteroid, or mesalamines after the qualifying endoscopy/radiology procedure up to randomization is permitted. Dose de-escalation after qualifying procedure is permissible at the discretion of the treating provider.
5. In corticosteroid-free symptomatic remission based on validated PROs (PRO2 score) and deemed to be experiencing no other IBD-related symptoms in the opinion of the treating provider. Includes patients who may be in medically induced remission (on index TIM); or surgically induced remission with post-op initiation of index TIM for prophylaxis and colonoscopy/imaging performed at least 3 months after initiation/optimization of TIM showing moderate-severe bowel inflammation. Validated PROs are defined as:

   1. CD: PRO2 (2-item patient reported outcome) mean daily score of abdominal pain score ≤1 and stool frequency score ≤ 3; or
   2. UC: PRO2, with absence of rectal bleeding (rectal bleeding score = 0) and with stool frequency score ≤1.
6. Evidence of moderate to severe bowel inflammation on local reading of colonoscopy, flexible sigmoidoscopy, balloon-assisted enteroscopy, capsule endoscopy or MR, CT enterography, or intestinal ultrasound, performed within 6 months prior to screening, defined at the investigator's discretion or as follows:

   1. CD: Colonoscopy showing moderately to severely active inflammation based on 1 of the following variables/scores:

      * Simple Endoscopic Score for Crohn's Disease (SES-CD) score ≥7 or score ≥4 for those with isolated ileal disease, or
      * Presence of mucosal ulcers >5 mm in size if SES-CD has not been recorded, or
      * Simplified Endoscopic Mucosal Assessment for Crohn's Disease (SEMA-CD) score ≥2, or
      * Rutgeerts score i2b or higher for patients in surgically induced remission with post-operative endoscopic recurrence [Note, either SES-CD or Rutgeerts score can be used for participants with post-operative recurrence]; or
   2. CD: MRE or CTE showing moderately to severely active inflammation based on 1 of the following variables:

      * Increased bowel wall thickness, or
      * Mural hyperenhancement, or
      * Peri-enteric fat stranding, or
      * Radiographic features of ulceration, or
      * Intramural T2 signal on fat suppressed images; or
   3. CD: Capsule endoscopy showing moderately to severely active small bowel disease based on Lewis score >790 (in case the disease is not accessible via endoscopy), or per local endoscopist if Lewis score is not reported; or
   4. CD: Gastrointestinal ultrasound showing at least 1 of the following variables:

      * Increased bowel wall thickness >5 mm, or
      * Color doppler score >5/cm2, or
      * Bowel stenosis, or
      * Bowel stratification, or
      * Fatty wrapping; or
   5. UC: modified MES score of 2 to 3, or documentation of any endoscopic feature that would define an MES of 2 to 3 (e.g., friability, ulceration, spontaneous bleeding, complete loss of vascular pattern), if an MES has not been recorded.
7. Eligible to receive at least 1 alternative TIM (excluding their index TIM) for the treatment of their disease per approved drug label, based on clinical and reimbursement guidelines.
8. Able to participate fully in all aspects of this clinical trial.
9. Informed consent must be obtained and documented.

EXCLUSION CRITERIA:

1. Presence of ostomy or ileoanal pouches.
2. Serious underlying disease other than UC or CD that in the opinion of the investigator may interfere with the participant's ability to participate fully in the study.
3. History of alcohol or drug abuse or any other medical or health condition that in the opinion of the investigator may interfere with the participant's ability to comply with the study procedures.
4. Prior enrolment in the current study.
5. Mild endoscopic disease activity, where treating providers would not consider switching TIM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Time to Treatment Failure | From randomization up to 104 weeks
  Time to treatment failure, as a composite of: (1) moderate severe symptomatic relapse based on PRO2, with objective confirmation of inflammation within 2 months of event (FC >250 mcg/g, or CRP >5mg/L, or endoscopy showing moderate-severe inflammation, or MRE/CTE/IUS showing active inflammation) with need for escalation of therapy; (2) need for rescue therapy with corticosteroids for a documented symptomatic IBD flare; (3) IBD related hospitalization; (4) IBD-related surgery; (5) IBD-related structural complications (CD: symptomatic stricture, fistula or abscess; UC: symptomatic stricture); (6) treatment-emergent adverse event requiring drug discontinuation

SECONDARY OUTCOMES:
Treatment failure as defined in the composite primary outcome | Binary, 104 weeks
  Treatment failure as defined in the composite primary outcome
Time to each individual component of the composite primary outcome | From randomization up to 104 weeks
  Time to each individual component of the composite primary outcome
Overall Quality of Life | Continuous, until 104 weeks or Early Discontinuation
  A) Scores of the SIBDQ. B) Scores of the IBD-Control. C) Scores of the PROMIS 7 scale. D) Scores of the on IBD-DI.
Treatment Burden/Satisfaction | Continuous, until 104 weeks or Early Discontinuation
  A) Scores of Treatment Burden Questionnaire, including medication, time and administrative, lifestyle change, social life and financial burden.
  B) Scores of Treatment Satisfaction Questionnaire for Medication, measuring treatment satisfaction across domains of effectiveness, side effects, convenience and global satisfaction.
  C) Scores of the CoPaQ, including out-of-pocket costs, for management of IBD, including treatment, monitoring, outpatient visits, and any unplanned healthcare utilization.
Overall Safety | Continuous, until 104 weeks or Early Discontinuation
  A) Treatment-related serious adverse events (SAEs) or unexpected SAEs. B) Serious infections, defined as infections requiring hospitalization and/or intravenous antibiotics.

CONTACTS AND LOCATIONS:
Overall Officials: Siddharth Singh, MD, Principal Investigator — UC San Diego Health
Locations (22):
- United States (22):
  - Hoag Hospital, Irvine, California
  - UC San Diego Health, La Jolla, California
  - Cedars-Sinai, Los Angeles, California
  - Sutter Health, Palo Alto, California
  - University of Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Chicago Medicine, Chicago, Illinois
  - Dartmouth Hitchcock, Lebanon, New Hampshire
  - Saratoga Schenectady Gastroenterology Associates, Burnt Hills, New York
  - NYU Langone Health, New York, New York
  - Cornell University, New York, New York
  - University of Rochester, Rochester, New York
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Oregon Clinic, Portland, Oregon
  - Gastroenterology Associates, Providence, Rhode Island
  - GastroOne, Germantown, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Utah Health, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh S, Nguyen JD, Fudman DI, Gerich ME, Shah SA, Hudesman D, McConnell RA, Lukin DJ, Flynn AD, Hwang C, Sprung B, Gaidos JKJ, Mattar MC, Rubin DT, Hashash JG, Metwally M, Ali T, Ma C, Hoentjen F, Narula N, Bessissow T, Rosenfeld G, McCurdy JD, Ananthakrishnan AN, Cross RK, Rodriguez Gaytan JR, Gurrola ES, Patel S, Siegel CA, Melmed GY, Weaver SA, Power S, Zou G, Jairath V, Hou JK. Treat-to-target of endoscopic remission in patients with inflammatory bowel disease in symptomatic remission on advanced therapies (QUOTIENT): rationale, design and protocol for an open-label, multicentre, pragmatic, randomised controlled trial. BMJ Open Gastroenterol. 2025 Mar 31;12(1):e001615. doi: 10.1136/bmjgast-2024-001615. PMID 40164445